CLINICAL TRIAL: NCT06945003
Title: Evaluating the Effectiveness of an Individualised Physical Activity Plan to Increase Exercise Capacity and Physical Activity Levels in Children With Congenital Heart Disease: A Randomised Control Trial
Brief Title: Study of Exercise Capacity and Physical Activity in Children With Congenital Heart Disease
Acronym: SHAPE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulster (Other)
Collaborators: Belfast Health and Social Care Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 322580
Record Dates: First submitted 2025-04-09; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Congenital Heart Disease
Keywords: children; adolescents; congenital heart disease; physical activity; exercise capacity
MeSH Terms: conditions — Heart Defects, Congenital; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Other): Those randomised to the control trial will be instructed to maintain their normal physical activity behaviours.
  If a participant is part of the control group, they will not receive the individualised physical activity plan, however their role is still very valuable. Control groups allow us as researchers to see if our 12-week individualised physical activity plan is effective at increasing exercise capacity and physical activity levels among children and adolescents with congenital heart disease. This information will help inform research and information given to families of children and adolescents with congenital heart disease in the future. At the end of the intervention, participants will be emailed the pre-recorded videos led by the fitness instructor demonstrating short games and activities that can be done as a family at home, that are fun and safe for children with congenital heart disease.
  Interventions: Behavioral: Exercise Intervention
- Intervention Group (Experimental): Those assigned to the intervention group will be invited to attend one of three group activity sessions with their parent/guardian that will occur at one of Ulster University's sport centres. Three group activity sessions will be delivered separately for each cohort (i.e Primary, Post-Primary and those with an Intellectual Disability) and their respective parent/guardian.) Parents/guardians and their child will then meet one-to-one with Professor Frank Casey, a paediatric cardiologist, will discuss with them, their child's results from their cardiopulmonary exercise test and from wearing their activity monitor. Using these results, alongside their age and diagnosis and likes and dislikes, Professor Casey will provide an individualised physical activity recommendation plan for each child that will be safe and beneficial to them, to be implemented at home over 12-weeks.
  Interventions: Behavioral: Exercise Intervention

INTERVENTIONS:
Behavioral: Exercise Intervention — Those assigned to the intervention group will be invited to attend one of three group activity sessions with their parent/guardian that will occur at one of Ulster University's sport centres. Three group activity sessions will be delivered separately for each cohort (i.e Primary, Post-Primary and those with an Intellectual Disability) and their respective parent/guardian.) Parents/guardians and their child will then meet one-to-one with Professor Frank Casey, a paediatric cardiologist, will discuss with them, their child's results from their cardiopulmonary exercise test and from wearing their activity monitor. Using these results, alongside their age and diagnosis and likes and dislikes, Professor Casey will provide an individualised physical activity recommendation plan for each child that will be safe and beneficial to them, to be implemented at home over 12-weeks.
  Other Names: SHAPE

SUMMARY:
Congenital heart disease (CHD) is the most common birth defect worldwide and occurs in every 8-10 per 1000 live births in Northern Ireland. The ability to participate in physical activity (PA) is an important aspect to an individual's quality of life. The UK Chief Medical Officer currently recommends that children aged 5-18 years should aim to achieve a minimum of 60 minutes PA per day. However, in Northern Ireland, only 8% of children with CHD are meeting these guidelines. This may be attributed to parents not allowing their child to fully participate in PA due to anxiety regarding its effect on their child's condition. Whilst, several studies to date have investigated the concerns faced by parents/guardians, this study is novel in its inclusion of teachers/coaches. Therefore, the investigators conducted interviews with parents/guardians and teachers/coaches to identify their concerns, highlighting that an individualised PA plan would help alleviate these fears.

This has informed a PA intervention, whereby the intervention group will receive an individualised PA plan to implement at home over a 12 week period with a 3 and 6 month follow up. This plan will also be sent out to teachers/coaches to inform them of what PA is both safe and beneficial for each child. The PA plan is adapted specifically for each child to increase their exercise capacity as this will increase their cardiorespiratory function and health related quality of life. It is also anticipated that it will increase PA level, thus increasing the percentage of children with CHD meeting current PA guidelines.

Therefore, the overall aim of this randomised control trial (RCT) is to assess the effectiveness of an individualised PA programme on exercise capacity and PA levels in children and adolescents with CHD. This will be assessed using both qualitative and quantitative methods.

DETAILED DESCRIPTION:
WHY THIS RESEARCH MATTERS The ability to take part in PA is an important aspect to an individual's quality of life. The UK Chief Medical Officer currently recommends that children aged 5-18 years should aim to be active for at least 60 minutes per day, however in Northern Ireland, only 13% of children are meeting these guidelines. This is worrying, as children with CHD are less active than healthy children, and it has been observed that children with complex CHD such as Fontan patients are less physically active than those with moderate CHD and their exercise capacity can be as low as 60% of reference value and further declines in adolescence and adulthood. This may be due to parents not allowing their child to fully participate in PA due to worries about their child's condition and non-cardiac comorbidities such as intellectual disabilities. Studies have suggested that parents of children with CHD are often apprehensive about their child's participation in PA, as a focus group study reported that parents and siblings often discouraged PA within the home, despite no clinical recommendation to do so. This study hypothesized that similarly, to parents, teachers and coaches may be apprehensive and unsure of the child's capabilities. However, no study to date has spoken to parents/guardians and teachers/coaches to investigate concerns faced regarding PA in children with CHD. Therefore, the investigators have conducted interviews with parents/guardians and teachers/coaches as in order to develop an effective and sustainable intervention, it is important to identify and address the concerns faced from those in the home and school environment who can either encourage or discourage PA among this population (Bagley et al. 2016; Ten Velde et al. 2021).

Previous studies have explored the effects of an individualised PA plan within children (5-10 years) and adolescents (12-20 years) however studies have shown that children are less active when they go to secondary school as PE lessons start to include more competitive sports (Callaghan et al. 2021; Morrison et al. 2013). Yet, no study to date has included all school-aged children (5-18 years) to identify if there are differences in PA levels when children transition from primary to secondary school.

In addition, children with intellectual disabilities such as those with Down Syndrome have been excluded from previous studies, even though they are less active than their peers. Therefore, this study will include all school aged children with CHD and an intellectual disability to participate in a PA intervention which will involve a PA plan, specific to each child, to be implemented at home. It is hypothesized that this study will improve PA levels and exercise capacity which will improve the child's health related quality of life.

This study is novel as it conducted qualitative interviews to inform an intervention that will be acceptable to the target population as parents/guardians and teachers/coaches have stated they would appreciate tailored PA as they highlighted that PA is not routinely discussed at appointments, despite the fact that relevant bodies published a statement recommending that encouraging daily participation in appropriate PA among children and adults should be a part of each patient encounter. Therefore, the investigators will develop an individualized home-based PA plan, with the aim of improving exercise capacity and PA levels which will in turn improve the child's health related quality of life and prognosis.

WHO WILL IT HELP There is currently no provision for individualized PA plans among this population despite recommendations from relevant bodies and qualitative interview feedback. Therefore this low-cost intervention aims to address this. By participating in this study, parents/guardians, children with CHD and teachers/coaches will have the opportunity to be provided with tailored PA and exercise recommendations on what is appropriate for them. This aims to reduce any anxiety parents/guardians, the children, and teachers/coaches may have about their participation in PA/exercise. PA can help improve children with congenital heart disease overall health, by improving their strength, muscle mass, reducing their risk of obesity and type 2 diabetes. PA can also help improve symptoms of anxiety and depression and overall quality of life and improve academic performance. Furthermore, the knowledge gained from this research will help improve the information and services surrounding physical activity provided to children with congenital heart disease and their families in the future.

The content and process of the programme incorporates features associated with effective interventions e.g. it is theory based; family centered; intervention was informed by parents/guardians and teachers/coaches who can either encourage or discourage among this population; uses evidence-based strategies and skilled staff who work consistently with this population.

The theories underpinning this PA programme are COM-B Model of Behaviour and the Self-Determination Theory.

Whilst sharing key characteristics of previous studies, it differs as it has been informed by qualitative interviews with parents/guardians and teachers/coaches to develop an intervention acceptable to those who can either encourage or discourage PA among this population. It is the first study to include all school-aged children to identify any changes in exercise capacity and PA levels between primary and post-primary school, when PA levels tend to decline. This is important to observe as sedentary behavior in adolescence often tracks into adulthood which is a risk factor for comorbidities such as obesity and type 2 diabetes. It is also the first study to include children and adolescents with an intellectual disability, which is vital as this population have the lowest PA levels. This study is also novel as the individualized PA plan, given the parent/guardian's consent will be posted to each child's teacher/coach to inform them of the child's condition and PA capabilities, including signs and symptoms to watch out for during PA.

Furthermore, this study will assess exercise capacity using cardiopulmonary exercise testing, which is a standard diagnostic test used among frequently among this population and is the gold-standard, however this was not used within previous studies.

Parents have also highlighted they feel their child would benefit from a visual aid such as a pre-recorded video. Therefore, we have identified a qualified sports development officer and fitness instructor with experience working with this population. The expert will pre-record a video demonstrating short games and activities that can be carried out at home with friends or family that are suitable and inclusive of this population.

Finally, a closed Facebook group will be created for participants >13 years and parents/guardians. The majority of those aged between 12-15 years own their own smartphone and have the highest rates of online activity compared to other populations. Facebook has been selected as it allows for a private group to be created that can be monitored and moderated by the researchers. It will be moderated by establishing clear rules and expectations for the group which will be displayed within the group description and as a welcome message. It will be monitored continuously by the PhD Researcher who will monitor and respond to posts and comments regularly. The PhD Researcher will review pending posts and check the group regularly for any inappropriate or spam content. Furthermore, a closed Facebook group allows the researchers to cross-check the participants age prior to accepting their request to join the group and only members can view who is in the group and their posts. This closed group will be used by the researcher to post encouraging messages about PA and the benefits of PA. It may also act as a prompt for participants and their parents/guardians to engage with the intervention. Finally, participants/parents/guardians can use the group to ask any questions they may have, post about upcoming PA activities or events that others may be interested in and to share their progress with their peers. This is novel as social media was not utilized within the previous studies, despite it's popularity with adolescents and adults.

THE INFORMATION THAT THIS STUDY WILL PROVIDE The proposed study will assess the effectiveness of an individualized PA plan for children and adolescents to increase exercise capacity, the percentage of those meeting PA guidelines, moderate to vigorous PA levels and health related quality of life. If effective, this PA programme could be easily implemented by paediatric cardiologists as it is low-cost and self-sustaining.

ELIGIBILITY:
Inclusion Criteria:

* Children with congenital heart disease aged 5-18 years (all diagnoses).
* Children with congenital heart disease aged 5-18 years and an intellectual disability.

Exclusion Criteria:

* Children or parents/guardians who do not wish to give assent or consent to participate in this study.
* Children with an underlying health condition and or physical disability in addition to congenital heart disease, to minimize the risk of confounding variables.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Exercise Capacity | 9 months
  The primary outcome measure will be exercise capacity to measure cardiorespiratory function among this population. Exercise capacity will be assessed by cardiopulmonary exercise testing (C-PET) to assess the individual's ability to exercise and the response of the individual's heart, lungs and muscles to exercise. C-PET remains the gold standard when assessing the functional limitations of cardiac patient and is a standard, low-risk, non-invasive, diagnostic test frequently used among this population and has been frequently used within intellectual disability populations.
  This will be performed on either a cycle ergometer or treadmill and will be conducted by a qualified cardiac physiologist in the presence of a paediatric cardiologist at RBHSC.

SECONDARY OUTCOMES:
Physical Activity Levels | 9 months
  Objectively measured total minutes moderate-to-vigorous physical activity (PA) will be measured using the GENEActive worn for 7 consecutive days.
  The device is wrist worn and participants will be asked to wear this device at all times over the 7-day period removing it only before bed. Tri-axial accelerometers such as the GENEActive device allow PA counts to be recorded in three dimensions and have been shown to be a valid measure of PA in children and adolescents.
Weight Measurements | 9 months
  Weight will be measured in kilograms (kg) to the nearest 0.1 kg using digital scales by a researcher trained in anthropometric techniques.
Height Measurements | 9 months
  Height will be measured in centimeters (cm) to the nearest 0.1 cm using a free-standing stadiometer.
Body Mass Index | 9 months
  Weight and height will be combined to report body mass index in kg/m^2
Waist Circumference | 9 months
  Waist circumference will be measured in centimeters (cm) to the nearest 0.1cm, using an anatomical measuring tape.
Hip Circumference | 9 months
  Hip circumference will be measured in centimeters (cm) to the nearest 0.1cm, using an anatomical measuring tape.
Waist-to-hip ratio | 9 months
  The waist measurement will be divided by the hip measurement to calculate waist-to-hip ratio.
Body Compostion | 9 months
  Body composition will be assessed using bioelectrical impedance analysis scales.
Health Related Quality of Life (HRQOL) | 9 months
  HRQOL will be assessed using The KIDSCREEN child self-report and parent proxy-report 27-item scale often used to assess HRQOL in children and adolescents with chronic health conditions. Parents of participants aged 5-7 years, will be asked to proxy report their child's HRQOL as the KIDSCREEN 27 is designed for children aged 8-18 years. Each item is measured on a 5-point response scale.

CONTACTS AND LOCATIONS:
Overall Officials: Professor Casey, Principal Investigator — Ulster University
Locations (1):
- Royal Belfast Hospital for Sick Children, Belfast, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared following the completion of this study due to confidentiality agreements with participants, institutional policies regarding data protection, and resource limitations that would be required for proper de-identification and data curation. The study team remains committed to research transparency through the publication of aggregate results and relevant statistical analyses while prioritizing participant privacy and adhering to all applicable data protection regulations.

REFERENCES:
- [Background] Teixeira PJ, Carraca EV, Markland D, Silva MN, Ryan RM. Exercise, physical activity, and self-determination theory: a systematic review. Int J Behav Nutr Phys Act. 2012 Jun 22;9:78. doi: 10.1186/1479-5868-9-78. PMID 22726453
- [Background] Stuart G, Forsythe L. Exercise prescription in young children with congenital heart disease: time for a change in culture. Open Heart. 2021 Jun;8(1):e001669. doi: 10.1136/openhrt-2021-001669. No abstract available. PMID 34083390
- [Background] Sparacino PS, Tong EM, Messias DK, Foote D, Chesla CA, Gilliss CL. The dilemmas of parents of adolescents and young adults with congenital heart disease. Heart Lung. 1997 May-Jun;26(3):187-95. doi: 10.1016/s0147-9563(97)90055-8. PMID 9176686
- [Background] Morrison ML, Sands AJ, McCusker CG, McKeown PP, McMahon M, Gordon J, Grant B, Craig BG, Casey FA. Exercise training improves activity in adolescents with congenital heart disease. Heart. 2013 Aug;99(15):1122-8. doi: 10.1136/heartjnl-2013-303849. Epub 2013 Jun 7. PMID 23749780
- [Background] Moola F, Faulkner GE, Kirsh JA, Kilburn J. Physical activity and sport participation in youth with congenital heart disease: perceptions of children and parents. Adapt Phys Activ Q. 2008 Jan;25(1):49-70. doi: 10.1123/apaq.25.1.49. PMID 18209244
- [Background] Michie S, van Stralen MM, West R. The behaviour change wheel: a new method for characterising and designing behaviour change interventions. Implement Sci. 2011 Apr 23;6:42. doi: 10.1186/1748-5908-6-42. PMID 21513547
- [Background] Matza LS, Swensen AR, Flood EM, Secnik K, Leidy NK. Assessment of health-related quality of life in children: a review of conceptual, methodological, and regulatory issues. Value Health. 2004 Jan-Feb;7(1):79-92. doi: 10.1111/j.1524-4733.2004.71273.x. PMID 14720133
- [Background] Longmuir PE, Corey M, McCrindle BW. Interactions with Home and Health Environments Discourage Physical Activity: Reports from Children with Complex Congenital Heart Disease and Their Parents. Int J Environ Res Public Health. 2021 May 4;18(9):4903. doi: 10.3390/ijerph18094903. PMID 34064527
- [Background] Kenzik KM, Tuli SY, Revicki DA, Shenkman EA, Huang IC. Comparison of 4 Pediatric Health-Related Quality-of-Life Instruments: A Study on a Medicaid Population. Med Decis Making. 2014 Jul;34(5):590-602. doi: 10.1177/0272989X14529846. Epub 2014 Apr 16. PMID 24739533
- [Background] Hinckson EA, Curtis A. Measuring physical activity in children and youth living with intellectual disabilities: a systematic review. Res Dev Disabil. 2013 Jan;34(1):72-86. doi: 10.1016/j.ridd.2012.07.022. Epub 2012 Aug 30. PMID 22940161
- [Background] Department of Health, 2019. Start active, stay active: a report on physical activity from the four home countries. Chief Medical Officers, London.
- [Background] Connolly S, Carlin A, Johnston A, Woods C, Powell C, Belton S, O'Brien W, Saunders J, Duff C, Farmer O, Murphy M. Physical Activity, Sport and Physical Education in Northern Ireland School Children: A Cross-Sectional Study. Int J Environ Res Public Health. 2020 Sep 19;17(18):6849. doi: 10.3390/ijerph17186849. PMID 32961784
- [Background] Callaghan S, Morrison ML, McKeown PP, Tennyson C, Sands AJ, McCrossan B, Grant B, Craig BG, Casey FA. Exercise prescription improves exercise tolerance in young children with CHD: a randomised clinical trial. Open Heart. 2021 May;8(1):e001599. doi: 10.1136/openhrt-2021-001599. PMID 33990433
- [Background] Blanchard J, McCrindle BW, Longmuir PE. The Impact of Physical Activity Restrictions on Health-Related Fitness in Children with Congenital Heart Disease. Int J Environ Res Public Health. 2022 Apr 7;19(8):4426. doi: 10.3390/ijerph19084426. PMID 35457294